CLINICAL TRIAL: NCT01168661
Title: Yoga, Mindfulness and Cognitive Psychotherapy as Treatment for Stress and Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Astrid Grensman, MD, Karolinska Institutet, Center for Family and Community Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pickup 2003
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Stress, Psychological; Burnout, Professional; Anxiety; Depression
Keywords: Stress; Burnout; Anxiety; Depression
MeSH Terms: conditions — Stress, Psychological; Burnout, Professional; Anxiety Disorders; Depression; Burnout, Psychological | interventions — Yoga; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control arm (No Intervention): Participants in this arm will be recruited from the group who applied to participate in the study and fulfilled the inclusion criteria but for various reasons (such as time constraints) could not participate.
- Cognitive psychotherapy arm (Active Comparator): In this arm, participants will attend a group meeting to practice cognitive psychotherapy once a week. They will also practice on their own >= 4 times a week.
  Interventions: Behavioral: Cognitive psychotherapy
- Mindfulness based cog psychotherapy arm (Active Comparator): In this arm, participants will attend a group meeting to practice mindfulness based cognitive psychotherapy once a week. They will also practice on their own >= 4 times a week.
  Interventions: Behavioral: Mindfulness based cog psychotherapy
- Yoga treatment group (Active Comparator): Persons in this arm will practice yoga >= 5 time each week (2 times in a supervised group and the other times on their own).
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Participants in this intervention arm will practice yoga (physical postures, breathing exercises, and meditation) >= 5 times a week (twice in a supervised group and the rest on their own). Additionally, participants in this arm will practice various practical skills, such as how to plan a satisfactory day using their own definition of a satisfactory day. They will follow this schedule for 20 weeks.
  Arms: Yoga treatment group
Behavioral: Mindfulness based cog psychotherapy — Participants in this arm will attend a weekly group meeting to practice mindfulness based cognitive psychotherapy. They will also practice >= 4 time a week on their own. Additionally, participants in this arm will practice various practical skills, such as how to plan a satisfactory day using their own definition of a satisfactory day. Participants will follow this schedule for 20 weeks.
  Arms: Mindfulness based cog psychotherapy arm
Behavioral: Cognitive psychotherapy — Participants in this arm will attend a weekly group meeting to practice cognitive psychotherapy. They will also practice >= 4 time a week on their own. Additionally, participants in this arm will practice various practical skills, such as how to plan a satisfactory day using their own definition of a satisfactory day. Participants will follow this schedule for 20 weeks.
  Arms: Cognitive psychotherapy arm

SUMMARY:
The purpose of this study is to investigate if treatment with yoga or mindfulness has a more profound and longstanding effect on stress and burnout than treatment with cognitive psychotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* On sick leave at least 50% at the beginning of the study.
* Sick leave for a maximum of 1 year if on full-time sick leave at the beginning of the study or for a maximum of 3 years if on part-time sick leave at the beginning of the study.
* Speak Swedish well enough to participate in the study interventions.
* Body mass index (BMI) of between 18 and 30.
* Meet the diagnostic criteria for burnout syndrome from the Swedish National Board of Health and Welfare.

Exclusion Criteria:

* Medication, including all medication or topical skin preparations with cortisone in any form. Exceptions: Antidepressants, contraceptives, hormone replacement therapy for hypothyroidism if hormone levels were within the normal range, and hormone replacement therapy to treat menopausal symptoms. To receive an exception for medication, a participant had to take the same medication at the same dose at both blood tests.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Reduced stress measured by qualitative questionnaires | 5 months after start of treatment
  Level of stress will be measured by qualitiative questionnaries, including the Swedish Health-Related Quality of Life Survey (SWEQUAL).

SECONDARY OUTCOMES:
Reduced cortisol secretion | 5 months after start of treatment
  We will measure cortisol level in a 24-hour sample of urine.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid M Grensman, MD, Principal Investigator — Karolinska Institutet; Bikash Dev Acharya, MSc Psyc, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Huddinge, Sweden

REFERENCES:
- [Derived] Grensman A, Acharya BD, Wandell P, Nilsson GH, Falkenberg T, Sundin O, Werner S. Effect of traditional yoga, mindfulness-based cognitive therapy, and cognitive behavioral therapy, on health related quality of life: a randomized controlled trial on patients on sick leave because of burnout. BMC Complement Altern Med. 2018 Mar 6;18(1):80. doi: 10.1186/s12906-018-2141-9. PMID 29510704